CLINICAL TRIAL: NCT05275881
Title: Impact of Virtual Reality in Hematology and Oncology for the Management of Pain During Invasive Procedures in Children, Adolescents and Young Adults, 7 to Under 25 Years in a Pilot Study
Brief Title: Impact of Virtual Reality in Hematology and Oncology During Invasive Procedures in Children, Adolescents and Young Adults, from 7 to Less Than 25 Years Old
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HOPPIVR
Record Dates: First submitted 2022-02-10; First posted 2022-03-11 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Virtual Reality; Pediatrics; Cancer; Pain; Procedural Pain
Keywords: Virtual Reality; Pediatrics; Cancerology; Pain; Invasive Acts
MeSH Terms: conditions — Neoplasms; Pain; Pain, Procedural

STUDY DESIGN:
Intervention Model Description: This is an exploratory interventional, comparative, single-center, randomized research into 2 parallel groups. The study will compare the use of virtual reality versus usual practices for two iterative and painful acts: lumbar puncture and connection to an implantable chamber.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality headset Group (Experimental): 30 patients will be included in the virtual reality arm
  Interventions: Device: Virtual Reality
- Control group with usual practices (Active Comparator): 30 patients will be included the usual practices
  Interventions: Drug: Usual Practices

INTERVENTIONS:
Device: Virtual Reality — In each arm, patients will benefit from an EMLA-type local anesthetic cream, pain and anxiety assessment. During the act, the physiological constants will be recorded (Fr, O2 and pulse). In the the RV group, The session will be started before the gesture and the patient will wear the helmet throughout the act. In case of pain and / or restlessness, the child will receive analgesics.
  Arms: Virtual Reality headset Group
Drug: Usual Practices — In each arm, patients will benefit from an EMLA-type local anesthetic cream, pain and anxiety assessment. During the act, the physiological constants will be recorded (Fr, O2 and pulse). In the control group, the child will receive the usual care: nitrous oxide, anxiolytics, opioid analgesics, psychotropic and benzodiazepine
  Arms: Control group with usual practices

SUMMARY:
This pilot study will be testing the feasibility of medical hypnosis through virtual reality during invasive médical procédures in children and young adults with cancer. Patients age from 7 to under 25 years whose treatement protocols required a lumbure puncture and a chemotherapy by implantable venous access will be randomly assigned to virtual reality or treatement as usual (nitrous oxide, anxiolytics, opioid analgesics, psychotropic and benzodiazepine). We expect the same benefit by using VR as usual intervention.

DETAILED DESCRIPTION:
Nationally, around 2,150 new cases of cancer are diagnosed per year in children aged 0 to 18. The main locations are leukemia, central system tumors and lymphomas. The onco-pediatrics unit of the Poitiers University Hospital is recruiting around 70 patients per year from 0 to under 18 years old. 1482 invasive procedures have been done in 2019. The diagnostic and therapeutic methods for these children remain aggressive and involve patients in chronic care. They repeatedly undergo painful and anxiety-inducing care. In pediatrics, nitrous oxide is chosen as the first-line choice in these various procedures, but its effectiveness is not always conclusive, due to habituation, and can induce side effects. For some children, it becomes difficult to obtain their consent to care, despite the range of different analgesics offered, and forces prescribers to increase the drugs. Virtual reality (VR) has already been shown to be effective on pain and anxiety in children and adolescents. This devices uses distraction and hypnosis techniques by establishing a state of hypnosedation and mediation through the work of breathing and sophrology. With this study, we expect the same benefit by using VR as usual pratices.

After explaining the treatment protocol, the potentially eligible patient will be informed by the investigator of the possibility of participating in this clinical trial. After checking the eligibility criteria and including the patient, the investigator can randomize the patient in the control group or the experimental group. As part of this study, patients will be followed for 1 month and for each act of lumbar puncture and connection to an implantable chamber.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 7 to strictly under 25
* Follow-ups for hematological or oncological pathology
* With a lumbar puncture or to connection to an implantable chamber
* Patient understanding French
* Consent of parents or guardians with parental authority.
* Child informed and having given his assent

Exclusion Criteria:

* Children with cognitive impairment
* Children in absolute emergency situations
* Children with a contraindication to a virtual reality headset (psychiatric pathology, vestibular and proprioceptive disorders, unbalanced epilepsy, impaired vision, hearing aids, claustrophobia, recent lesions of the eyes, face or scalp)
* Children who have already participated in the clinical investigation
* Refusal to participate in the study
* Patients not benefiting from a social security system or not benefiting from it by the intermediary of a third person

Ages: 7 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-11-13 (Estimated); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of virtual reality compared to usual analgesic practices in pain management during the first lumbar puncture or connection to an implantable chamber of the study. | up to one day
  At the inclusion, the primary endpoint will be to assess pain using the Visual Analogue Scale (VAS) after the first invasive act of lumbar puncture or connection to an implantable chamber.
  The pain assessment will be carried out using a Visual Analogue Scale provided as part of the clinical investigation.The EVA (Analogue Visual Assessment) from 0 to 10, is a scale that can be used from the age of 7. It reliably allows self-assessment of pain.
  The scale will be explained to the child before the act and it will be presented to him after the invasive act for the assessment:
  * 0: no pain
  * Between 1 and 3: mild pain
  * Between 3 and 5: moderate-intensity pain
  * Between 5 and 7: severe pain
  * Greater than 7: very intense pain

SECONDARY OUTCOMES:
Comparison, between the control group and the group supported with virtual reality: Pain from the VAS after the 1st connection to the implantable chamber | up to one month
  Pain from the VAS after the 1st connection to the implantable chamber:
  The pain assessment will be carried out using a Visual Analogue Scale provided as part of the clinical investigation.The VAS (Visual Analogue Assessment) from 0 to 10, is a scale that can be used from the age of 7. It reliably allows self-assessment of pain.
  The scale will be explained to the child before the act and it will be presented to him after the invasive act for the assessment:
  * 0: no pain
  * Between 1 and 3: mild pain
  * Between 3 and 5: moderate-intensity pain
  * Between 5 and 7: severe pain
  * Greater than 7: very intense pain
Comparison, between the control group and the group supported with virtual reality: Child's anxiety using the Frankl scale | up to one month
  The Frankl scale, is a scale of hetero-evaluation of anxiety. It will be performed by the caregiver before the invasive procedure (lumbar puncture and connection to an implantable chamber). It is suitable for children from 7 to under 25 years old and is easy to score:
  * 0: Definitely negative behavior; refuses treatment, shouts forcefully, opposes/cares,
  * 1: Negative behavior: unwilling to accept care; unwilling to accept care. Some signs of opposition exist but not necessarily declared (sullen air, scowling),
  * 2: Positive behaviour; accepts treatment with reservation. He is cautious but follows the instructions of the practitioner/caregiver
  * 3: Definitely positive behavior; good relations/practitioner/caregiver, interested in treatment. He laughs often and seems to enjoy the visit/care.
Comparison, between the control group and the group supported with virtual reality:The type and amount of analgesics consumed during the invasive act (lumbar puncture and / or connection to an implantable chamber) | up to one month
  The type of associated analgesics, the dosage will be collected through the patient's medical record
Comparison, between the control group and the group supported with virtual reality: Heart rate | up to one month
  Heart rate (min <40 B/min - max >200 B/min), from a scope connected to the patient before and throughout the duration of the invasive act (lumbar puncture and / or connection to an implantable chamber)
Comparison, between the control group and the group supported with virtual reality:oxygen saturation | up to one month
  oxygen saturation (min <90% - max >100%) from a scope connected to the patient before and throughout the duration of the invasive act (lumbar puncture and / or connection to an implantable chamber)
Comparison, between the control group and the group supported with virtual reality: Respiratory rate | up to one month
  Respiratory rate (min <10 - max > 50) from a scope connected to the patient before and throughout the duration of the invasive act (lumbar puncture and / or connection to an implantable chamber)
Comparison, between the control group and the group supported with virtual reality: Tolerance | up to one month
  Tolerance, in number of episodes of confusion, agitation, dizziness, nausea, vomiting, headache, hallucinations and temporary amnesia during the performance of the invasive act and within 2 hours of post-act monitoring for a lumbar puncture and 30 minutes for a connection to an implantable chamber
Comparison, between the control group and the group supported with virtual reality: Pain after each act from the VAS | up to one month
  A patient may have several consecutive invasive acts. The pain assessment will be carried out using a Visual Analogue Scale provided as part of the clinical investigation.The VAS (Visual Analogue Assessment) from 0 to 10, is a scale that can be used from the age of 7:
  * 0: no pain
  * Between 1 and 3: mild pain
  * Between 3 and 5: moderate-intensity pain
  * Between 5 and 7: severe pain
  * Greater than 7: very intense pain
Comparison, between the control group and the group supported with virtual reality: Pain from the VAS after the 1st connection to an implantable chamber | up to one month
  Pain from the VAS after the 1st connection to an implantable chamber the :
  The pain assessment will be carried out using a Visual Analogue Scale provided as part of the clinical investigation.The VAS (Visual Analogue Assessment) from 0 to 10, is a scale that can be used from the age of 7. It reliably allows self-assessment of pain.
  The scale will be explained to the child before the act and it will be presented to him after the invasive act for the assessment:
  * 0: no pain
  * Between 1 and 3: mild pain
  * Between 3 and 5: moderate-intensity pain
  * Between 5 and 7: severe pain
  * Greater than 7: very intense pain

CONTACTS AND LOCATIONS:
Overall Officials: Amandine AF FERNANDES, Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No